CLINICAL TRIAL: NCT03534947
Title: A Pilot Study to Evaluate Short Term Neoadjuvant Sonidegib Followed by Surgery or Imiquimod in the Management of Basal Cell Carcinomas in Cosmetically Challenging Locations
Brief Title: A Study to Evaluate Neoadjuvant Sonidegib Followed by Surgery or Imiquimod in the Management of Basal Cell Carcinoma
Acronym: SONIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIA2017/CT/220; HREC file number 18/087 (Other: Human Research Ethics Committee)
Record Dates: First submitted 2018-05-01; First posted 2018-05-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Basal Cell Carcinoma; Basal Cell Carcinoma of Skin, Site Unspecified; Skin Cancer; Invasive Carcinoma
Keywords: Neoadjuvant; Sonidegib
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — sonidegib; Imiquimod; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This is a pilot study which will evaluate the efficacy and safety of short term neoadjuvant sonidegib followed by surgery or imiquimod in the management of basal cell carcinomas in cosmetically challenging locations, assessed by optical coherence tomography and histopathology. The data from this pilot study may lead to the design of larger scale trials of neoadjuvant targeted therapy with the aim to decrease the morbidity of surgical treatment and increase the probability of a curative resection in larger patient populations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sonidegib followed by imiquimod (Experimental): Sonidegib 200mg taken orally once a day for 12 weeks. COMPLETE OR PARTIAL RESPONSE WITH SUPERFICAL REMNANT LESION For patients with a complete response or a partial response resulting in a superficial lesion, treatment with topical imiquimod for 5 days a week for 6 weeks will be prescribed.
  Interventions: Drug: Sonidegib; Drug: Imiquimod
- Sonidegib followed by surgery (Experimental): Sonidegib 200mg taken orally once a day for 12 weeks. PARTIAL RESPONSE WITH REMNANT INVASIVE LESION For patients with a no change on BCC size / depth or patients with a partial response but a remaining invasive lesion, will have surgical excscion of the remaining lesion.
  Interventions: Drug: Sonidegib; Procedure: Surgery
- Sonidegib then best supportive care (Other): Sonidegib 200mg taken orally once a day for 12 weeks. PROGRESSIVE DISEASE Patients with lesions that have progressed in size and/or depth will receive the best supportive care deemed appropriate by the treating clinician. This may be surgery, imiquimod, a clinical trial treatment, radiotherapy or any combination of these interventions.
  Interventions: Drug: Sonidegib; Other: Best supportive care

INTERVENTIONS:
Drug: Sonidegib — Sonidegib is a selective and orally bioavailable Smoothened (Smo) antagonist. The dose will be 200mg taken once a day for 12 weeks.
  Other Names: LDE225; Odomzo
Drug: Imiquimod — Imiquimod is an immune response modifier that promotes NF-kappa-B-mediated secretion of pro-inflammatory cytokines, chemokines and other mediators. These immune responses produce cytotoxic effects that are antiproliferative and anti-tumour. Imiquimod treatment requires an extended treatment period of 6 weeks for superficial BCC. Imiquimod is an option for the treatment of small, low-risk superficial BCC when surgery, curettage or cryotherapy are inappropriate. Treatment with imiquimod will be for 5 days a week for a total of 6 weeks.
  Other Names: Aldara
  Arms: Sonidegib followed by imiquimod
Procedure: Surgery — Although most BCCs are amenable to surgery, excision of large tumours in aesthetically sensitive sites may compromise function or cosmesis. Patients whose BCC has not shrunk in size or depth following 12 weeks of sonidegib will undergo surgical excision of the remaining tumour.
  Other Names: Excision of remnant invasive basal cell carcinoma
  Arms: Sonidegib followed by surgery
Other: Best supportive care — Patients with lesions that have progressed in size and/or depth will receive the best supportive care deemed appropriate by the treating clinician. This may be surgery, imiquimod, a clinical trial treatment, radiotherapy or any combination of these interventions
  Arms: Sonidegib then best supportive care

SUMMARY:
In this study, patients with BCC will be given neoadjuvant treatment with a drug called sonidegib. Sonidegib is a daily tablet usually given for BCC that cannot be removed by surgery or that has spread through the body. The study aims to see if sonidegib given for 12 weeks will reduce the size of tumours so surgery results in less scarring or may be avoided, with only short term topical treatment required to treat remaining tumour.

DETAILED DESCRIPTION:
Surgery is the first line treatment for most basal cell carcinomas (BCCs) with cure rates of 88 to 96%. However, excision of large lesions in sensitive locations such as the face and scalp may result in disfigurement and impairment of function. Neoadjuvant drug treatment given before surgery aims to reduce tumour size so that surgery and recovery is easier. In this study, patients with BCC will be given neoadjuvant treatment with a drug called sonidegib. Sonidegib is a daily tablet usually given for BCC that cannot be removed by surgery or that has spread through the body. The study aims to see if sonidegib given for 12 weeks will reduce the size of tumours so surgery results in less scarring or may be avoided, with only short term topical treatment required to treat remaining tumour. This approach may also reduce the risk of recurrence. To assess response to treatment, we will use a new technology for skin tumours called optical coherence technology (OCT). This is like an ultrasound scan and is non invasive. OCT can detect the extent and nature of the tumour and build a 3D image with great accuracy. OCT will be used together with pathological analysis of tumour tissue to determine response to sonidegib.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Written informed consent.
* Histologically confirmed, resectable, invasive basal cell carcinoma.
* Site and size of BCC considered to be in a cosmetically challenging position for surgery.
* Patient has expressed concerns of the cosmetic outcome of surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Ability to swallow and retain oral medication.
* Anticipated life expectancy of > 12 months.
* Adequate organ function as demonstrated by blood tests.
* Willing to abstain from blood donations for 20 months from the last dose of sonidegib.
* Men with female partner of childbearing potential to use effective contraception from 14 days prior to study treatment until 6 months after the last dose.
* Female patients with active contraception or no menstrual cycle for >12 months

Exclusion Criteria:

* Inoperable basal cell carcinoma tumours.
* A concurrent cancer diagnosis requiring any systemic anti-cancer therapy.
* Serious or unstable pre-existing medical conditions or other conditions or laboratory abnormalities that could interfere with the patient's safety, consent, or compliance.
* History of malabsorption or other conditions that would interfere with the absorption of sonidegib.
* Known psychiatric or substance abuse disorders that would interfere with cooperation and compliance with the requirements of the trial.
* Prior treatment with hedgehog pathway inhibitors.
* Concomitant medications that may result in increased or decreased bioavailability of sonidegib.
* Patients with neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, rhabdomyolysis, amyotrophic lateral sclerosis and spinal muscular atrophy) due to an increased risk of muscle toxicity with sonidegib.
* Male patients expecting to father children or donate sperm during the 12 weeks of sonidegib treatment and for a further 6 months from the end of treatment.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Neoadjuvant treatment response determined by optical coherence tomography | 12 weeks
  The size and spread of abnormal skin structures associated with basal cell carcinoma detected by optical coherence tomography.

SECONDARY OUTCOMES:
Neoadjuvant treatment response determined by histopathology | 12 weeks
  The size and spread of basal cell carcinoma tumour in a biopsy taken from the known worse affected area of disease demonstrated by histopathologic analysis.
Histologic response to neoadjuvant treatment in basal cell carcinoma sub types | 12 weeks
  The amount and spread of basal cell carcinoma tumour cells and structures detected at histopathology analysis in nodular and in infiltrative sub types of BCC.
Response to neoadjuvant treatment in basal cell carcinoma sub types measured with optical coherence tomography. | 12 weeks
  The amount and spread of basal cell carcinoma tumour cells and structures detected at histopathology analysis in nodular and in infiltrative sub types of BCC.
Recurrence rate | 6 and 12 months after surgery or at the end of 6 weeks of treatment with imiquimiod.
  The number of patients who have a recurrence of basal cell carcinoma at the original site of disease after having surgery or 6 weeks of topical treatment with imiquimod.
Drug related adverse reactions | 12 weeks
  The proportion of patients experiencing any adverse drug reactions graded according to CTCAE version 4.
Discontinuation of sonidegib due to adverse reactions | 12 weeks
  The proportion of patients who discontinue sonideigb because of adverse drug reactions.
Quality of life based on SKINDEX-16 | Weeks 12 and 18 and months 6 and 12.
  The scores obtained from the validated SKINDEX-16 quality of life questionnaire compared to baseline.
Patient rated cosmetic outcome after neoadjuvant treatment followed by surgery | Week 12
  Scores from a 3 likert scale questions assessing the patient's agreement with statements about the appearance of their surgical scar for patients who need surgery after neoadjuvant treatment.
Surgeon rated cosmetic outcome after neoadjuvant treatment followed by surgery | Week 12
  Scores from a 3 likert scale questions assessing the surgeon's agreement with statements about the appearance of their surgical scar for patients who need surgery after neoadjuvant treatment.
Patient rated cosmetic outcome after neoadjuvant treatment | Week 12
  Scores from a 3 likert scale questions assessing the patient's agreement with statements about the appearance of the remmant BCC area for patients who did not need surgery after neoadjuvant treatment.
Surgeon rated cosmetic outcome after neoadjuvant treatment | Week 12
  Scores from a 3 likert scale questions assessing the surgeons's agreement with statements about the appearance of the remmant BCC area for patients who did not need surgery after neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Guitera, MD PhD, Study Director — Melanoma Institute Australia
Locations (1):
- Melanoma Institute Australia, North Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang AL, Atwood SX, Tartar DM, Oro AE. Surgical excision after neoadjuvant therapy with vismodegib for a locally advanced basal cell carcinoma and resistant basal carcinomas in Gorlin syndrome. JAMA Dermatol. 2013 May;149(5):639-41. doi: 10.1001/jamadermatol.2013.30. No abstract available. PMID 23677114
- [Background] Cheng HM, Guitera P. Systematic review of optical coherence tomography usage in the diagnosis and management of basal cell carcinoma. Br J Dermatol. 2015 Dec;173(6):1371-80. doi: 10.1111/bjd.14042. Epub 2015 Oct 27. PMID 26211438
- [Background] Cheng HM, Lo S, Scolyer R, Meekings A, Carlos G, Guitera P. Accuracy of optical coherence tomography for the diagnosis of superficial basal cell carcinoma: a prospective, consecutive, cohort study of 168 cases. Br J Dermatol. 2016 Dec;175(6):1290-1300. doi: 10.1111/bjd.14714. Epub 2016 Sep 24. PMID 27146027
- [Background] Ching JA, Curtis HL, Braue JA, Kudchadkar RR, Mendoza TI, Messina JL, Cruse CW, Smith DJ Jr, Harrington MA. The impact of neoadjuvant hedgehog inhibitor therapy on the surgical treatment of extensive basal cell carcinoma. Ann Plast Surg. 2015 Jun;74 Suppl 4:S193-7. doi: 10.1097/SAP.0000000000000452. PMID 25695449